CLINICAL TRIAL: NCT01626807
Title: Evaluation of a Walking School Bus Program: A Cluster Randomized Controlled Trial
Brief Title: Evaluation of a Walking School Bus Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Jason Mendoza, Associate Professor of Pediatrics, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R01CA163146-01A1 (NIH)
Record Dates: First submitted 2012-06-21; First posted 2012-06-25 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Obesity; Physical Activity
Keywords: Safe Routes to School; Walking School Bus; Cluster Randomized Controlled Trial; Physical Activity; Obesity; Overweight
MeSH Terms: conditions — Obesity; Motor Activity; Overweight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Walking school bus (Experimental)
  Interventions: Behavioral: Walking School Bus
- Usual care (No Intervention)

INTERVENTIONS:
Behavioral: Walking School Bus — Children will have the option of walking to and/or from school with study staff who are trained in Safe Routes to School methods.
  Arms: Walking school bus

SUMMARY:
Just two generations ago, walking or bicycling to school was the norm for a substantial number of US children, e.g. 48% of children walked or biked to school in 1969 versus only 13% in 2009. This decline occurred in the same timeframe as the childhood obesity epidemic, which is at record high levels in the US and affects low-income and ethnic minority children the most. This project will test "the walking school bus" (WSB) program, in which children walk to and from school with adults, and its impact on low-income, ethnic minority children's walking to school, physical activity, and risk for obesity. Ultimately, this line of research has the potential to provide a low-cost, easy to disseminate program to reduce risk of obesity and cancer for at-risk children.

The investigators Specific Aims among 3rd-5th grade children include:

SA1) To recruit 770 child-parent dyads from 22 elementary schools over 4 years and conduct a cluster randomized controlled trial to assess the efficacy of a WSB program on children's walking to school, physical activity, and BMI z-score over a school-year SA2) To collect and analyze data on individual-, school-, and macro-level influences on changes to children's walking to school resulting from the WSB program

The Primary Hypotheses to be tested, in comparison to control children, include:

H1) The WSB program will increase children's walking to school over a school-year.

H1a) Parents' outcome expectations and self-efficacy will mediate the relationship between the WSB and changes to children's walking to school.

H1b) Walkability, safety, and acculturation will moderate changes to children's walking to school.

H2) The WSB program will increase children's physical activity and decrease BMI z-scores over a school-year.

H3) The WSB program will increase school-level pedestrian safety behaviors over a school-year.

ELIGIBILITY:
Inclusion Criteria:

* physically capable of walking to and from school
* live within 1-mile of school or parents agree to regularly drop off children within 1-mile of school
* attend a study school and enrolled in 3rd, 4th, or 5th grade

Exclusion Criteria:

* another child from the same household is enrolled in the study

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 838 (Actual)
Dates: Start 2012-12; Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Weekly rate of children's active commuting to school | 5-6 months

SECONDARY OUTCOMES:
Moderate-to-vigorous physical activity | 5-6 months
Body mass index z-score | 5-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jason A Mendoza, MD, MPH, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Research Institute, Seattle, Washington, United States

REFERENCES:
- [Derived] Johnson AM, Zhou C, Haviland M, Mendoza JA. Evaluation of a walking school bus program: a cluster randomized controlled trial. Int J Behav Nutr Phys Act. 2024 May 10;21(1):55. doi: 10.1186/s12966-024-01602-w. PMID 38730407
- See also: Walking School Bus Guidelines — http://guide.saferoutesinfo.org/walking_school_bus/index.cfm